CLINICAL TRIAL: NCT01184118
Title: Does Inhaled Fluticasone REsult in Obstructive Sleep Apnea? DREAM-A Pilot Study
Brief Title: DREAM: Does Inhaled Fluticasone REsult in Obstructive Sleep Apnea Manifestations?
Acronym: DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Brigham and Women's Hospital (Other); University of California, San Diego (Other); University of California, San Francisco (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2008-0265; U10HL074212 (NIH)
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-07

CONDITIONS: Lung Disease
Keywords: asthma; sleep apnea
MeSH Terms: conditions — Lung Diseases; Asthma; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FP Discontinued (No Intervention): The design is a prospective 16-week open-label study of inhaled FP hydrofluoroalkane-propelled metered dose inhaler (HFA-MDI), 220 mcg, 4 puffs BID in 36 ICS naive asthma subjects. This is followed by a 4-week run-out period, including FP 220 mcg 2 puffs BID for 2 weeks, then either continue FP 220 mcg 2 puffs BID or discontinue FP (as tolerated), for the remaining two weeks, with subsequent transition to clinical care.
- FP 220 mcg 2 puffs BID (Active Comparator): The design is a prospective 16-week open-label study of inhaled FP hydrofluoroalkane-propelled metered dose inhaler (HFA-MDI), 220 mcg, 4 puffs BID in 36 ICS naive asthma subjects. This is followed by a 4-week run-out period, including FP 220 mcg 2 puffs BID for 2 weeks, then either continue FP 220 mcg 2 puffs BID or discontinue FP (as tolerated), for the remaining two weeks, with subsequent transition to clinical care.
  Interventions: Drug: FP 220 mcg 2 puffs BID

INTERVENTIONS:
Drug: FP 220 mcg 2 puffs BID — The design is a prospective 16-week open-label study of inhaled FP hydrofluoroalkane-propelled metered dose inhaler (HFA-MDI), 220 mcg, 4 puffs BID in 36 ICS naive asthma subjects. This is followed by a 4-week run-out period, including FP 220 mcg 2 puffs BID for 2 weeks, then either continue FP 220 mcg 2 puffs BID or discontinue FP (as tolerated), for the remaining two weeks, with subsequent transition to clinical care.
  Other Names: Fluticasone propriante
  Arms: FP 220 mcg 2 puffs BID

SUMMARY:
This study is being conducted to find out if the use of inhaled corticosteroids has an affect on upper airway (UAW) collapsibility and sleep apnea risk. An inhaled corticosteroid is a common asthma controller medication like Flovent. Sleep apnea or sleep deprived breathing (SDB) is when someone stops breathing for a short period of time during sleep. For some reason, people with asthma have more sleep apnea and upper airway (UAW) collapsibility (weakness) than the general population. There are many possible reasons for this and one might be related to the use of inhaled corticosteroids.

The overall hypothesis of this study is to determine whether inhaled fluticasone propionate (FP) increases UAW collapsibility and to assess tongue (genioglossus muscle) dysfunction as a potential underlying mechanism.

DETAILED DESCRIPTION:
To address this hypothesis, we specifically aim is to determine the effects of 16 weeks of treatment with inhaled FP hydrofluoroalkane-propelled metered dose inhaler (HFA-MDI), 880 mcg twice daily, on:

Specific Aim 1: UAW collapsibility, as measured by Pcrit during NREM sleep; Specific Aim 2: Severity of obstructive SDB and sleep quality, and quality of life related to sleep apnea assessed on validated questionnaires (Sleep Apnea scale of the Sleep Disorders Questionnaire [SA-SDQ], Epworth Sleepiness Scale [ESS]) and Pittsburgh Sleep Quality Index [PSQI], and Sleep Apnea Quality of Life Index [SAQLI]); Specific Aim 3: Tongue strength and fatigability (assessed using the Iowa Oral Performance Instrument)

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65;
2. history consistent with asthma
3. symptoms consistent with NAEPP26 asthma severity step ≥2 (in the past 2-4 weeks, presence of any of the following: daytime symptoms >2 days/week; or nighttime symptoms 3-4x/month; or short acting bronchodilator use (not for prevention of exercise induced asthma) >2 days/week, requiring addition on a controller therapy, using the NAEPP Asthma Step Categorization guidelines
4. FEV1≥65%
5. confirmation of asthma diagnosis by bronchodilator reversibility (≥12% improvement in FEV1 from baseline following 2 puffs of a β-2 agonist) or a provocative concentration of methacholine needed to produce a 20% fall in FEV1 (PC20) of ≤ 8 mg/ml.

Exclusion Criteria:

1. any use of inhaled corticosteroid for >2 weeks at a time during the last 6 months, or any use in the last 6 weeks
2. as needed use of nasal steroids in the prior 6 months (regular use is allowed without washout needed prior to testing visits)
3. use of medications listed in Table 1. Inhaled long acting β-adrenergics are permitted for entry and should be continued during this study
4. respiratory infection during the prior 4 weeks or asthma exacerbation during the prior 6 weeks to enrollment
5. presence of other lung diseases
6. evidence of significant medical (such as angina, heart failure, stroke) or psychiatric illnesses
7. diagnosed osteopenia (on treatment) or osteoporosis
8. established diagnosis of neuromuscular disease (e.g. multiple sclerosis, syringomyelia, transverse myelitis, amyotrophic lateral sclerosis (ALS), poliomyelitis, Lambert Eaton syndrome, Guillain-Barre syndrome, myasthenia gravis, myotonic dystrophy, mononeuritis multiplex, in the setting of polymyositis/dermatomyositis or severe cervical spine disease)
9. BMI greater than 35 kg/m2
10. currently on treatment for OSA
11. new diagnosis of OSA if OAI > 10/hour or desaturation <70% on dPSG (V2
12. pregnancy or desire to get pregnant in the upcoming 6 months (subjects of child-bearing potential must agree to use an acceptable method of birth control per ACRN guidelines, as stated in the consent form: i.e. if not post-menopausal [1 year or more since last menses] or surgically sterile [hysterectomy, tubal ligation, or vasectomy in monogamous partner], subject must use one of the following acceptable birth control methods: abstinence, birth control pills, diaphragm, intra-uterine device [IUD], Norplant, Depo-Provera, NuvaRing, birth control patches [e.g., Ortho Evra], single or double barrier methods [condom plus foam/jelly or condom plus diaphragm])
13. cigarettes > 1pack/month or cigars in the year before study or overall tobacco use greater than 10 pack years
14. inability to abstain from alcohol ingestion for 24 hours prior to sleep studies
15. any current use of benzodiazepins, opioids or barbiturates; 16) any current use of recreational drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Teodorescu, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Univeristy of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- FP 220 mcg 2 Puffs BID: The design is a prospective 16-week open-label study of inhaled FP hydrofluoroalkane-propelled metered dose inhaler (HFA-MDI), 220 mcg, 4 puffs BID in 36 ICS naive asthma subjects. This is followed by 2 weeks of FP 220 mcg 2 puffs BID then either continue FP 220 mcg 2 puffs BID or discontinue FP (as tolerated), for the remaining two weeks.
Period: Overall Study
Arm/Group | FP 220 mcg 2 Puffs BID
Started | 36
FP MDI 1,760 mcg/Day (16 Weeks) | 18
FP MDI 880 mcg/Day (2 Weeks) | 18
FP MDI as Indicated (2 Weeks) | 18
Completed | 18
Not Completed | 18
Not completed — Only asthma step 1 - screen fail | 1
Not completed — No physiologic confirmation of asthma | 8
Not completed — FEV1 <60% predicted | 2
Not completed — Exclusionary medical condition | 2
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | FP 220 mcg 2 Puffs BID
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved, Unchanged, and Worsened Critical Closing Pressure (Pcrit) From Baseline With 16-week of High Dose Inhaled FP Treatment.
Description: Upper airway (UAW) collapsibility, as measured by critical closing pressure (Pcrit), defined as the maximum nasal pressure at which the UAW occludes. Subjects were divided into 3 subgroups: improved (more negative Pcrit), unchanged, or worsened (less negative Pcrit).
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | FP 220 mcg 2 Puffs BID
Number analyzed (Participants) | 18
participants
  Improved Pcrit over 16 weeks | 8
  Unchanged Pcrit over 16 weeks | 8
  Worsened Pcrit over 16 weeks | 2

2. Secondary Outcome: Number of Participants With Improved, Unchanged, and Worsened Sleep Disorders Questionnaire (SA-SDQ) From Baseline With 16-week of High Dose Inhaled FP Treatment.
Description: Secondary goals include evaluating effects of this medication on severity of obstructive sleep disordered breathing (SDB) (validated by Sleep Disorders Questionnaire (SA-SDQ)). Subjects were divided into 3 subgroups: improved (less negative SA-SDQ score), unchanged, or worsened (more negative SA-SDQ score).
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | FP 220 mcg 2 Puffs BID
Number analyzed (Participants) | 18
participants
  Improved SA-SDQ score over 16 weeks | 8
  Unchanged SA-SDQ score over 16 weeks | 8
  Worsened SA-SDQ score over 16 weeks | 2

3. Secondary Outcome: Number of Participants With Improved, Unchanged, and Worsened Anterior Tongue Strength (KPa) From Baseline With 16-week of High Dose Inhaled FP Treatment.
Description: The Iowa Oral Performance Instrument (IOPI) will be used. This instrument has a standard-sized air-filled polymer balloon, called tongue sensor or bulb, which can be inserted between the tongue blade and the roof of the mouth. Anterior tongue strength (KPa) reported. Subjects were divided into 3 subgroups: improved (lower anterior tongue strength KPa), unchanged, or worsened (higher anterior tongue strength KPa).
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | FP 220 mcg 2 Puffs BID
Number analyzed (Participants) | 18
participants
  Improved Anterior tongue strength over 16 weeks | 8
  Unchanged Anterior tongue strength over 16 week | 8
  Worsened Anterior tongue strength over 16 week | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 2 years.
Arm/Group | FP 220 mcg 2 Puffs BID
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

LIMITATIONS AND CAVEATS:
We were unsuccessful at securing placebo MDI, and the lack of a control group raises the possibility that our findings may reflect natural history of pharyngeal upper airway patency in asthma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No